CLINICAL TRIAL: NCT06559501
Title: Integrated Case Management for Improved Psychosocial and Physical Rehabilitation of Burn Survivors and Their Families Treated in Pakistan
Brief Title: Integrated Case Management for Burns Care in Pakistan
Acronym: BURNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PILL-BURNS-OO1
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Unintentional Burn Injury; Depression; Anxiety; Burns
Keywords: Burns Rehabilitation; culturally adapted; Cost effectiveness; Multicenter trial; Pakistan; Burns Injury
MeSH Terms: conditions — Depression; Anxiety Disorders; Burns

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated case manager care (Experimental): comprises 8 sessions delivered by case managers. Case managers will provide up to 6 low-intensity sessions in the hospital or the community (if the patient is discharged before completing the required sessions), with content and duration tailored to patient preferences. Post-discharge, patients will receive 2 follow-up sessions with case managers to ensure a smooth transition into the community.
  Interventions: Behavioral: Integrated case manager care
- Enhanced care as usual (No Intervention): includes their standard care, and all treatments recommended by attending physicians will be provided, plus a written self-help booklet

INTERVENTIONS:
Behavioral: Integrated case manager care — comprises 8 sessions delivered by case managers. Case managers will provide up to 6 low-intensity sessions in the hospital or the community (if the patient is discharged before completing the required sessions), with content and duration tailored to patient preferences. Post-discharge, patients will receive 2 follow-up sessions with case managers to ensure a smooth transition into the community.
  Arms: Integrated case manager care

SUMMARY:
To test whether a culturally adapted multicomponent intervention for improving burns care and patient/family rehabilitation is effective in improving survival among burn victims in Pakistan and is cost-effective. The comparator will be usual care plus brief written self-help advice (enhanced usual care). The study is designed as a multicentre, pragmatic, parallel group, individually randomised trial. Participants in the intervention arm will receive 8 sessions delivered by the case managers (6 low-intensity sessions lasting 30-60 minutes in the hospital/community and 2 follow-up sessions lasting 30 minutes in the community). Assessments will be conducted at baseline, at 3 months, 6 months and at 12-months post-intervention.

DETAILED DESCRIPTION:
The Burns trial will be conducted in six cities of Pakistan; Karachi, Hyderabad, Lahore, Rawalpindi, Peshawar and Quetta to compare integrated intervention with enhanced usual care. Participants will be randomized either to the intervention or enhanced usual care. The intervention consists of multiple culturally adapted components such as psychological bundle, emergency care, surgical and rehab bundle to improve care within burn units, transitional care, and patient and family rehabilitation (known as 'Integrated case management for improved psychosocial and physical rehabilitation of burn survivors and their families'). The comparator will be usual care (emergency, surgical and rehab care ) plus brief written self-help booklets will be given(enhanced usual care).

The intervention will be carried out by case managers (trained allied health professionals such as nurses, physiotherapists, psychologists etc) and will be started during hospital stay to enhance physical health outcomes by educating patients about self-care/ medications and adherence to treatment resources provided to the case managers and upon discharge to the participants and their carers.

Participants in the intervention arm will receive 8 sessions delivered by the case managers (6 low-intensity sessions lasting 30-60 minutes in the hospital/community and 2 follow-up sessions lasting 30 minutes in the community). Assessments will be conducted at baseline, at 3 months, 6 months and at 12-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and over
* Accidental burn injury and meet the criteria for admission to burn centres
* Clinician judgment for participation readiness
* Ability to provide informed consent

Exclusion Criteria:

No intentional burn injuries

• Lacking capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1146 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Hierarchical composite score of all-cause mortality, all cause hospital readmissions and health related quality of life (EQ5D) | Baseline to 12th month post randomization
  all-cause mortality followed by readmission rates and changes in health-related quality of life

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Baseline to 3 months, 6 months and 12-months post-intervention
  To screen, diagnose, monitor and measure the severity of depression
Burns Specific Health Scale | Baseline to 3 months, 6 months and 12-months post-intervention
  To quantify dysfunction and distress across six major domains of health, specifically burn injury related morbidity
Rosenburg Self-Esteem Scale | Baseline to 3 months, 6 months and 12-months post-intervention
  A 10 item self-report instrument to measure individual self-esteem
Visual Analogue Scale | Baseline to 3 months, 6 months and 12-months post-intervention
  It provides subjective magnitude estimation and consists of a straight line with limits that carry a verbal description of each extreme of the symptom both pain relief or pain severity
International Trauma Questionnaire | Baseline to 3 months, 6 months and 12-months post-intervention
  It is a brief,18 item self-report questionnaire used to assess core features of Post-Traumatic Stress Disorder (PTSD) and Complex PTSD.
Perceived Stigma Questionnaire | Baseline to 3 months, 6 months and 12-months post-intervention
  It is used to measure stigmatizing behaviors commonly reported by people with appearance distinctions. Participants were asked to rate how often they experienced a behavior on a 5-point Likert scale
WHO disability assessment schedule | Baseline to 3 months, 6 months and 12-months post-intervention
  It is used to measure the impact of health condition, functioning, disability, monitor the effectiveness of interventions as well as the burden of disease both mental and physical disorders
Vancouver Scar Scale | Baseline to 3 months, 6 months and 12-months post-intervention
  It is used to document change in scar appearance. Index measures the scares on four parameters, Pigmentation, vascularity, pliability and heigh
Quality of life scale EQ-5D | Baseline to 3 months, 6 months and 12-months post-intervention
  Health-related quality of life as measured for mobility, self-care, usual activities, pain/discomfort and anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, MD, Principal Investigator — Pakistan Institute of Living and Learning
Locations (11):
- Pakistan (11):
  - Burn Unit, Sandeman Provisional Hospital, Quetta, Balochistan
  - Plastic Surgery and Burn Unit, BMC, Quetta, Quetta, Balochistan
  - Burns and Plastic Surgery Center, Peshawar, Peshawar, KPK
  - Department of Plastic, Reconstructive Surgery and Burn Unit, Kind Edward Medical University, Lahore, Punjab Province
  - Jinnah Burn & Reconstructive Surgery Centre, Lahore, Lahore, Punjab Province
  - Pak Italian Modern Burn and Plastic Surgery Centre, Multan Khurd, Punjab Province
  - Burn Centre, Civil Hospital Hyderabad, Hyderābād, Sindh
  - Burn Centre, Ruth K. M. Pfau, Civil Hospital Karachi, Karachi, Sindh
  - Burns and Plastic Surgery, Patel Hospital, Karachi, Karachi, Sindh
  - Allied Burn & Reconstructive Surgery Centre, Faisalābad
  - Burn Care Centre, PIMS, Islamabad, Islamabad

IPD SHARING:
Plan to Share IPD: No
Available on reasonable request

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Blades B, Mellis N, Munster AM. A burn specific health scale. J Trauma. 1982 Oct;22(10):872-5. doi: 10.1097/00005373-198210000-00012. PMID 7131607
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Rosenberg M. Rosenberg self-esteem scale. Journal of Religion and Health. 1965
- [Background] Langley GB, Sheppeard H. The visual analogue scale: its use in pain measurement. Rheumatol Int. 1985;5(4):145-8. doi: 10.1007/BF00541514. PMID 4048757
- [Background] Cloitre M, Shevlin M, Brewin CR, Bisson JI, Roberts NP, Maercker A, Karatzias T, Hyland P. The International Trauma Questionnaire: development of a self-report measure of ICD-11 PTSD and complex PTSD. Acta Psychiatr Scand. 2018 Dec;138(6):536-546. doi: 10.1111/acps.12956. Epub 2018 Sep 3. PMID 30178492
- [Background] Lawrence JW, Fauerbach JA, Heinberg LJ, Doctor M, Thombs BD. The reliability and validity of the Perceived Stigmatization Questionnaire (PSQ) and the Social Comfort Questionnaire (SCQ) among an adult burn survivor sample. Psychol Assess. 2006 Mar;18(1):106-11. doi: 10.1037/1040-3590.18.1.106. PMID 16594819
- [Background] Üstün TB. Measuring health and disability: Manual for WHO disability assessment schedule WHODAS 2.0: World Health Organization; 2010.
- [Background] Baryza MJ, Baryza GA. The Vancouver Scar Scale: an administration tool and its interrater reliability. J Burn Care Rehabil. 1995 Sep-Oct;16(5):535-8. doi: 10.1097/00004630-199509000-00013. PMID 8537427